CLINICAL TRIAL: NCT04669587
Title: A Phase 1/2, Open-label, Multicenter Study to Evaluate the Safety, Tolerability, Preliminary Antitumor Activity, Pharmacokinetics, and Pharmacodynamics of ZB716 as Monotherapy and in Combination With Palbociclib in Patients With Estrogen Receptor-Positive, HER2-Negative Locally Advanced or Metastatic Breast Cancer
Brief Title: ER+/HER2- Locally Advanced or Metastatic Breast Cancer (ENZENO Study)
Acronym: ENZENO
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: EnhancedBio USA Inc. (Other)
Collaborators: Zenopharm (Unknown)
Responsible Party: Sponsor
Organization: EnhancedBio Inc. (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ENZENO-C-101
Record Dates: First submitted 2020-11-15; First posted 2020-12-17 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Estrogen Receptor-Positive; HER2-Negative; Locally Advanced Breast Cancer; Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — palbociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part A: Dose Escalation of ZB716 monotherapy (with Food Effect Cohort) (Experimental): Cohorts will follow a 3+3 study design. Approx. 3 to 6 subjects will be enrolled in each dose cohort (6 subjects in Cohort A6; food-effect evaluation). (Dose levels: 50, 100, 200, 300, 400 mg, orally QD in a 28 day cycle) The overall DLT observation period of ZB716 monotherapy will be 4 weeks following the initial dose of study drug on Cycle 1 Day 1. There will be 2 ~ 6 days between dose escalations to allow sufficient time for an adequate safety review. The max. dose may be lower than 400 mg. In the first dosing group of Part A (Cohort A1), subject dosing will be staggered such that administration of the first dose is separated by at least 7 days between the first 2 subjects. In each of Cohorts A1 to A5, 3 to 6 subjects will receive ZB716 doses according to the assigned dose level in the fasted state. For Cohort A6, Period 1, doses will be administered in the fasted state in Treatment Period 1 and 2, doses will be given 30 min. after starting a standard high fat breakfast.
  Interventions: Drug: ZB716
- Part B: Dose Expansion of ZB716 monotherapy (Experimental): Potential subjects will be screened to assess their eligibility to enter the study within 28 days prior to the first dose administration. Subjects will come to the clinical site before the first dose of study drug to confirm eligibility. Cohorts will be enrolled sequentially based on an optional Simon 2-stage study design.
  Approx. 29 subjects may be enrolled in the dose expansion cohorts of Part B. For Part B, doses will be administered (self-administered by subjects at home or administered by subjects under observation of clinical staff during clinic visits) at the determined monotherapy RD of ZB716 (based on Part A) QD in a 28-day cycle. Doses will be administered in the dietary status for dosing as determined from Part A fed/fasted comparison.
  Interventions: Drug: ZB716
- Part C: Dose Escalation of ZB716 in combination with palbociclib (Experimental): Cohorts will follow a 3+3 study design. Approx. 6 to 12 subjects will be enrolled in the dose escalation phase of ZB716 in combination with Palbociclib. For Part C, doses will be administered at escalating doses starting with 1 dose level below the monotherapy RD (determined in Part A) and Palbociclib will be dosed at the fixed standard dose of 125 mg QD. ZB716 will be administered on a 28 day cycle and Palbociclib will be administered for 21 days in the cycle with 7 days off treatment. Administration of the higher dose level (at monotherapy RD) of ZB716 (with the standard dose of Palbociclib) to subsequent subjects will be based on the occurrence of DLTs during the DLT observation period (Cycle 1), until MAD of ZB716 with combination of Palbociclib is reached. Doses will be administered in the dietary status for dosing as determined from Part A fed/fasted comparison.
  Interventions: Drug: ZB716; Drug: Palbociclib
- Part D: Dose Expansion of ZB716 in combination with palbociclib (Experimental): Potential subjects will be screened to assess their eligibility to enter the study within 28 days prior to the first dose administration. Subjects will come to the clinical site before the first dose of study drug to confirm eligibility. Cohorts will be enrolled sequentially based on an optional Simon 2-stage study design.
  Approx. 29 subjects may be enrolled in the dose expansion cohorts of Part D. For Part D, doses will be administered (self-administered by subjects at home or administered by subjects under observation of clinical staff during clinic visits) at the determined RD of ZB716 QD for 28 days from Part C in combination with the standard dose of Palbociclib (125 mg QD for 21 days with 7 days off treatment). Doses will be administered in the dietary status for dosing as determined from Part A fed/fasted comparison.
  Interventions: Drug: ZB716; Drug: Palbociclib

INTERVENTIONS:
Drug: ZB716 — Pharmaceutical form: capsule Route of administration: oral
  Other Names: Borestrant
Drug: Palbociclib — Pharmaceutical form: capsule Route of administration: oral
  Other Names: Ibrance®
  Arms: Part C: Dose Escalation of ZB716 in combination with palbociclib; Part D: Dose Expansion of ZB716 in combination with palbociclib

SUMMARY:
For patients with ER-positive, HER2-negative breast cancer, blockage of the ER pathway has been proven to be an effective anticancer approach. These patients showed good response to endocrine therapy.

Fulvestrant, the approved SERD as monotherapy or in combination with CDK4/6 inhibitors, showed superior clinical benefit compared to other endocrine therapies. Fulvestrant exhibits differential mechanism of action from other endocrine therapy, such as tamoxifen, aromatase inhibitors, which indicates that direct blockage of ER might derive better clinical activity.

However, due to its route of administration by intramuscular injection, the clinical application is limited, especially with long term use. In addition, a higher dose of fulvestrant at 500 mg showed better overall survival than the lower dose at 250 mg, suggesting that more profound ER pathway modulation could derive better clinical benefit. Therefore, a SERD with improved oral bioavailability and good safety profile which enables its overdose is anticipated to achieve a more satisfactory clinical outcome with better compliance of clinical use.

Preclinical data indicates that ZB716 is a novel orally bioavailable, selective ERα degrader with full ER antagonism that demonstrates superior properties than Fulvestrant. Thus, it has a potential to be effective therapy for patients with ER-positive breast cancer.

This is the first time ZB716 will be administered to humans. The principal aim of this study is to obtain safety and tolerability data when ZB716 is administered orally as monotherapy and in combination with palbociclib to subjects with ER-positive, HER2 negative advanced breast cancer. This information, together with the PK data, will help establish the doses and dosing regimen suitable for future studies in patients. The PD effect of ZB716 on the select biomarkers for cytochrome P450 (CYP)3A4 induction (4β hydroxycholesterol) and expression of ER, PgR, and Ki67 will also be investigated. The effect of ZB716 on antitumor activity as measured by objective response rate (ORR), clinical benefit rate (CBR), duration of response (DOR), and PFS rate will also be investigated. The study will also investigate the effects of food on the PK of ZB716 monotherapy.

ELIGIBILITY:
[Inclusion Criteria]

Subjects must satisfy all of the following criteria for study entry:

1. Subjects must be able to understand the nature of the trial and provide a signed and dated, written informed consent form (ICF) prior to any study-specific procedures, sampling, and analyses.
2. Subjects aged ≥18 years old at time of signing ICF (or country's legal age of majority if the legal age is >18 years).
3. Histologically or cytologically confirmed diagnosis of adenocarcinoma of the breast.
4. Subjects with evidence of either locally advanced disease not amenable to radiation therapy or surgery in a curative intent, or metastatic disease.
5. ER-positive tumor (≥1% positive stained cells) based on most recent tumor cell staining by immunohistochemistry (IHC) assay consistent with local standards.

Note: If primary tumor is ER-positive and any further metastatic lesions are ER negative, the subject cannot be selected for inclusion.

[Exclusion Criteria]

Subjects who meet any of the following criteria will be excluded from study entry:

1. Treatment with any systemic anticancer therapies for locally advanced or metastatic breast cancer within 4 weeks or 5 half-lives of prior anticancer therapy, whichever is shorter, prior to initiation of study treatment.
2. Concurrent treatment with warfarin or phenytoin.
3. Diagnosis of any secondary malignancy within 3 years prior to enrollment, except for all intraepithelial neoplasia, appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, or Stage I uterine cancer.
4. Active inflammatory bowel disease, chronic diarrhea, short bowel syndrome, major upper gastrointestinal (GI) surgery including gastric resection, or any other condition that may affect absorption of oral study drug.
5. Known clinically significant history of liver disease consistent with Child-Pugh Class B or C, including active viral or other hepatitis (eg, hepatitis B or hepatitis C virus), current alcohol abuse, or cirrhosis. Active viral or positive test for viral hepatitis as defined below:

Note: If reports of serology test for HBV and HCV containing normal ranges issued by formal medical institutions within 28 days prior to C1D1 (and prior to informed consent) are available, these tests are exempt while screening. Unless required by local regulations, patients are not required to have HIV assessments at screening.

Active infection is defined as requiring treatment with antiviral therapy or presence of positive test results for hepatitis B (hepatitis B surface antigen [HBsAg] and/or total hepatitis B core antibody [HBcAb]) or HCV antibody.

Patients who test positive for HBcAb are eligible only if test results are also positive for hepatitis B surface antibody and polymerase chain reaction is negative for HBV DNA.

Patients who are positive for HCV serology are only eligible if testing for HCV RNA is negative.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2021-07-26 (Actual); Primary Completion 2023-01-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Part A: To determine the RD(Recommended Dose) of ZB716 | At the end of Cycle 1 (each cycle is 28 days)
  Incidence of study treatment-related DLTs at Cycle 1
Part B: To assess antitumor activities at the ZB716 RD in monotherapy | Baseline to the date of first documentation of progression, assessed approximately up to 6 months after the last entered patient
  Proportion of patients with CR(Complete Response), PR(Partial Response) or SD(Stable Disease) according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 assessed by independent central reviewer relative to the total number of treated patients
Part C: To determine the RD of ZB716 in combination with palbociclib | At the end of Cycle 1 (each cycle is 28 days)
  Incidence of study treatment-related DLTs at Cycle 1
Part D: To assess antitumor activities in the combination therapy of ZB716 and Palbociclib | Baseline to the date of first documentation of progression, assessed approximately up to 6 months after the last entered patient
  Proportion of patients with CR(Complete Response), PR(Partial Response) or SD(Stable Disease) according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 assessed by independent central reviewer relative to the total number of treated patients

SECONDARY OUTCOMES:
Adverse Events (Part A, B, C and D) | Up to 30 days after last dose of ZB716 or ZB716 with Palbociclib
  Number of patients with adverse events according to the National Cancer Institute - Common Toxicity Criteria (NCI-CTC) version 5.0 grade scaling. Incidence of adverse events, including laboratory test results and electrocardiogram (ECG) findings that were adverse events
ORR(Object Response Rate) (Part A, B, C and D) | Baseline to the date of first documentation of progression, assessed approximately up to 6 months after the last entered patient
  Proportion of patients with CR(Complete Response) or PR(Partial Response) according to RECIST 1.1 assessed by investigator/local radiologist
CBR(Clinical Benefit Rate) (Part A and C) | Baseline to the date of first documentation of progression, assessed approximately up to 6 months after the last entered patient
  Proportion of patients with CR(Complete Response) or PR(Partial Response) or SD(Stable Disease) ≥16 weeks according to RECIST v.1.1 relative to the total number of treated patients by investigators/local radiologists
Duration of response (Part A, B, C and D) | Baseline to the date of first documentation of progression, assessed approximately up to 6 months after the last entered patient
  Time from initial response to the first documented tumor progression
Cmax of ZB716 after single dose (Part A, B, C and D) | Cycle 0, Day -7 (Part A), Cycle 1, Day 1 (Part B, C and D) (each cycle is 28 days)
  Cmax is maximum concentration observed.
Tmax of ZB716 after single dose (Part A, B, C and D) | Cycle 0, Day -7 (Part A), Cycle 1, Day 1 (Part B, C and D) (each cycle is 28 days)
  Tmax is time to reach Cmax.
AUC0-24 of ZB716 after single dose (Part A, B, C and D) | Cycle 0, Day -7 (Part A), Cycle 1, Day 1 (Part B, C and D) (each cycle is 28 days)
  AUC0-24 is area under the plasma concentration versus time curve calculated using the trapezoidal method over the dosing interval (24 hours)
Cmax of ZB716 after repeated dose (Part A, B, C and D) | Cycle 2, Day 1 (Part A), Cycle 1, Day 15 (Part B, C and D) (each cycle is 28 days)
  Cmax is maximum concentration observed.
Tmax of ZB716 after repeated dose (Part A, B, C and D) | Cycle 2, Day 1 (Part A), Cycle 1, Day 15 (Part B, C and D) (each cycle is 28 days)
  Tmax is time to reach Cmax.
AUC0-24 of ZB716 after repeated dose (Part A, B, C and D) | Cycle 2, Day 1 (Part A), Cycle 1, Day 15 (Part B, C and D) (each cycle is 28 days)
  AUC0-24 is area under the plasma concentration versus time curve calculated using the trapezoidal method over the dosing interval (24 hours)
Cmax of Palbociclib after single dose (Part C and D) | Cycle 1, Day 1 (Part C and D) (each cycle is 28 days)
  Cmax is maximum concentration observed.
Tmax of Palbociclib after single dose (Part C and D) | Cycle 1, Day 1 (Part C and D) (each cycle is 28 days)
  Tmax is time to reach Cmax.
AUC0-24 of Palbociclib after single dose (Part C and D) | Cycle 1, Day 1 (Part C and D) (each cycle is 28 days)
  AUC0-24 is area under the plasma concentration versus time curve calculated using the trapezoidal method over the dosing interval (24 hours)
Cmax of Palbociclib after repeated dose (Part C and D) | Cycle 1, Day 15 (Part C and D) (each cycle is 28 days)
  Cmax is maximum concentration observed.
Tmax of Palbociclib after repeated dose (Part C and D) | Cycle 1, Day 15 (Part C and D) (each cycle is 28 days)
  Tmax is time to reach Cmax.
AUC0-24 of Palbociclib after repeated dose (Part C and D) | Cycle 1, Day 15 (Part C and D) (each cycle is 28 days)
  AUC0-24 is area under the plasma concentration versus time curve calculated using the trapezoidal method over the dosing interval (24 hours)

CONTACTS AND LOCATIONS:
Locations (8):
- Swedish Cancer Institute, Seattle, Washington, United States
- South Korea (7):
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - CHA Bundang Medical Center, CHA University, Seongnam-si
  - Korea University Anam Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No